CLINICAL TRIAL: NCT06452862
Title: the Value of Multimodal Magnetic Resonance Imaging in the Diagnosis and Treatment Monitoring of Diabetic Kidney Disease
Brief Title: Multimodal Magnetic Resonance Imaging in Evaluation of Diabetic Kidney Disease
Status: Recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yu Shi, Deputy director of department of radiology, Shengjing Hospital
Other Study IDs: ShengjingH-DKD
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Kidney Disease
Keywords: Diabetic Kidney Disease; Magnetic Resonance Imaging; Magnetic Resonance Elastography; Diabetes
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetics: Participants with diagnosed Diabetes will undergo the same MRI protocol as the Healthy Volunteers, including Blood Oxygen Level Dependence (BOLD), Intravoxel Incoherent Motion (IVIM), Arterial Spin Labeling (ASL), T1&T2-mapping imaging and Magnetic Resonance Elastography (MRE). In addition to the imaging, these participants will have their blood creatinine, cystatin C, and blood pressure measured within 3 days before and after the MRE. A renal biopsy will be performed as part of their clinical assessment to evaluate the extent of kidney damage.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging
- Healthy Volunteers: Age-matched healthy individuals with no known kidney disease will be recruited. They will undergo the same MRI protocols as the Diabetics group, including Blood Oxygen Level Dependence (BOLD), Intravoxel Incoherent Motion (IVIM), Arterial Spin Labeling (ASL), T1&T2-mapping imaging and Magnetic Resonance Elastography (MRE), to establish baseline viscoelasticity parameters for comparison with the Diabetics.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Both Diabetics and Healthy Volunteers will undergo MRI protocols including Blood Oxygen Level Dependence (BOLD), Intravoxel Incoherent Motion (IVIM), Arterial Spin Labeling (ASL), T1&T2-mapping imaging and Magnetic Resonance Elastography (MRE). For Diabetics, blood tests for creatinine and cystatin C, along with blood pressure measurements, will be taken within a three-day window surrounding the MRE test. Additionally, Diabetics will undergo a renal biopsy to assess the extent of kidney damage.

SUMMARY:
The goal of this study is to investigate the value of noninvasive evaluation of multimodal magnetic resonance imaging in diagnosis and treatment of diabetic kidney disease (DKD). We aim to explore the feasibility of multimodal magnetic resonance imaging in the staging diagnosis of DKD, and establish a non-invasive method for evaluating the progression of DKD disease by combining imaging and biochemical indicators. Multimodal magnetic resonance examinations will be performed on diabetic patients with different stages as well as regular follow-up during treatment, in order to investigate the relationship between imaging findings and pathophysiological changes of the kidneys.

DETAILED DESCRIPTION:
At present, the clinical diagnosis of diabetic kidney disease (DKD) relies mainly on the detection of urine microalbumin，which is influenced by many other factors. Renal biopsy is another modality to detect DKD, but it cannot be widely used in clinical practice because of its invasiveness. Thus, a reproducible and reliable noninvasive method is needed for more accurate diagnosis.

Multimodal magnetic resonance imaging, which including but not limited to magnetic resonance elastography (MRE), blood oxygen level-dependent magnetic resonance imaging (BOLD-MRI), arterial spin labeling (ASL), incoherent motion diffusion-weighted imaging (IVIM-DWI), T1mapping and T2mapping, is able to provide valuable information about subtle structural and functional changes, and has shown promising potential in the diagnosis, classification and prediction of pathological and molecular features.

In this clinical trial, multimodal magnetic resonance examinations will be performed on diabetic patients with different stages as well as regular follow-up during treatment, in order to investigate the relationship between imaging findings and pathophysiological changes of the kidneys. We aim to explore the feasibility of multimodal magnetic resonance imaging in the staging diagnosis of DKD and establish a non-invasive method for evaluating the progression of DKD disease by combining imaging and biochemical indicators, in order to provide reference for clinical medication. This research could be helpful for better understanding and management of DKD, and pave the way for more accurate diagnosis, improved clinical decision-making, personalized treatment approaches for DKD patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed diabetes
* No other diseases that affect renal function (such as gout, blood related diseases, primary hypertension, nephrotic syndrome, etc.),
* No contraindications for magnetic resonance imaging examination

Exclusion Criteria:

* Image quality does not meet the measurement requirements.
* Renal function damage caused by non-diabetes factors
* Combined with other important organ dysfunction
* Combined with malignant tumor
* Combined with other metabolic diseases anemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subject inclusion criteria were adult patients with diabetes without non-diabetic kidney injury.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Imaging Evaluation of Kidney | Baseline to 6 months
  To evaluate the ability of Multimodal Magnetic Resonance Imaging to identify and quantify the extent of of kidney damage. Regions of interest (ROIs) were placed manually in the renal cortex and medulla, avoiding renal hilar vessels and areas of obvious artifacts.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Shi, M.D., Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown RS, Sun MRM, Stillman IE, Russell TL, Rosas SE, Wei JL. The utility of magnetic resonance imaging for noninvasive evaluation of diabetic nephropathy. Nephrol Dial Transplant. 2020 Jun 1;35(6):970-978. doi: 10.1093/ndt/gfz066. PMID 31329940